CLINICAL TRIAL: NCT07364812
Title: The Effect of Intraoperative Findings Shown to the Patient on Early Postoperative Clinical Outcomes in Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E.167479
Record Dates: First submitted 2025-04-30; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Arthroplasty Replacement, Knee; Gonarthrosis; Primary
Keywords: arthroplasty; knee; gonarthrosis; effect; photograph
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: After the surgery, when the patient was cooperative and open to communication, they were visited and informed that intraoperative photos were taken and could be shown to them if desired. Patients who wanted to see the photos were included in the study, while those who declined formed the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photo Group (Active Comparator): Patients who want to see intraoperative photos
  Interventions: Behavioral: The Effect of Showing Intraoperative Cartilage Damage and Post-Implantation Range of Motion Photos to Patients on Early Clinical and Functional Outcomes in Patients Undergoing Total Knee Arthroplasty
- Control Group (Placebo Comparator): The patients who dont want to see intraoperative photos and also after the patients in the first group are accumulated, all subsequent patients
  Interventions: Behavioral: The Effect of Showing Intraoperative Cartilage Damage and Post-Implantation Range of Motion Photos to Patients on Early Clinical and Functional Outcomes in Patients Undergoing Total Knee Arthroplasty

INTERVENTIONS:
Behavioral: The Effect of Showing Intraoperative Cartilage Damage and Post-Implantation Range of Motion Photos to Patients on Early Clinical and Functional Outcomes in Patients Undergoing Total Knee Arthroplasty — Before discharge, usually on the second day, active knee flexion and extension were noted while the patient was in the supine position. During the postoperative 2nd and 6th-week follow-up visits, the range of motion was also recorded.
  Preoperative VAS, Oxford Knee Score, SF-12 Physical, and SF-12 Mental scores were obtained from patients after admission. Additionally, the same scores were re-recorded during the 6-week follow-up visit.
  At the 6-week follow-up, patients underwent the Timed Up and Go (TUG) test, Stair Climb Test (SCT), and 6-minute walk tests, and their scores were recorded.

SUMMARY:
The Effect of Showing Intraoperative Cartilage Damage and Post-Implantation Range of Motion Photos to Patients on Early Clinical and Functional Outcomes in Patients Undergoing Total Knee Arthroplasty

Objective: The aim of this study is to determine the early clinical and functional effects of showing photos of intraoperative cartilage damage and range of motion after prosthetic implantation to patients who undergo Total Knee Arthroplasty as part of the treatment for advanced gonarthrosis (stage 3-4).

Patients and Methods: The study was initiated at Bezmialem Vakıf University with approval from the Ethics Committee (Approval Number: E.167479) on 03.10.2024. With a 95% confidence level and 80% power (average difference of 4 units, standard deviation of 6.3), at least 40 patients per group (2 groups) are required. Data will be analyzed using IBM SPSS Statistics 22.0 software. The t-test will be used to compare the mean differences of continuous variables between groups, the Chi-square test will be used for the distribution of categorical variables between groups, and Pearson correlation coefficient will be used to analyze the relationship between continuous variables. Descriptive statistics will include mean, standard deviation, correlation coefficient (r), frequency, and percentage values. A p-value of <0.05 will be considered statistically significant.

Exclusion criteria for our study include revision total knee arthroplasty surgeries, total knee arthroplasty surgeries following high tibial osteotomy, total knee arthroplasty surgeries after unicompartmental knee arthroplasty, and surgeries with advanced deformities requiring the use of revision implants.

DETAILED DESCRIPTION:
On the day of surgery, patients were examined in their preoperative beds while in the supine position, and knee flexion and extension were recorded. After the capsulotomy, the distal femoral cartilage surface defects were photographed. Additionally, after prosthetic implantation, photos of the prostheses were taken. After the surgery was completed and dressing was applied, the patient was asked to perform knee flexion and extension while lying in the supine position, and a photo was taken.

After the surgery, when the patient was cooperative and open to communication, they were visited and informed that intraoperative photos were available and could be shown if desired. Patients who wanted to see the photos were included in the study, while those who declined formed the control group. Patients were shown the defect in the cartilage of their knee and informed that after the prostheses were implanted, they would achieve full joint range of motion. It was advised that they mobilize more safely during postoperative rehabilitation.

Pre-discharge, usually on the second day, active knee flexion and extension were noted while the patient was in the supine position. During the postoperative 2nd and 6th-week follow-up visits, the range of motion was again recorded.

Assessment and Data Collection: Preoperative VAS, Oxford Knee Score, SF-12 Physical, and SF-12 Mental scores were obtained from patients after admission. These same scores were repeated and recorded during the 6-week follow-up visit.

At the 6-week follow-up, patients underwent the Timed Up and Go (TUG) test, Stair Climb Test (SCT), and 6-minute walk test, and their scores were recorded.

The collected data will be analyzed to determine the differences between the study group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone Total Knee Arthroplasty as part of the treatment for advanced gonarthrosis (stage 3-4)

Exclusion Criteria:

* Revision total knee arthroplasty surgeries
* total knee arthroplasty surgeries following high tibial osteotomy
* total knee arthroplasty surgeries following unicompartmental knee arthroplasty
* surgeries with advanced deformities requiring the use of revision implants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
VAS (Visual Analog Scale for Pain) | From preop to 6 weeks
  What is a VAS score?
  VAS stands for Visual Analog Scale. It's a simple way to measure how strong a feeling or symptom is, most often pain, but it can also be used for things like fatigue, stress, or nausea.
  How does the VAS work?
  The VAS is usually shown as a straight line.
  One end means "no pain" (or no symptom).
  The other end means "worst pain imaginable" (or the worst possible symptom).
  The person marks a point on the line that best matches how they feel.
  How is it scored?
  The line is usually 10 cm (100 mm) long.
  The score is measured from the "no pain" end to the mark.
  This gives a number:
  0 = no pain
  10 (or 100) = worst pain possible
Oxford Knee Score (OKS) | From preop to 6 weeks
  What is the Oxford Knee Score?
  The Oxford Knee Score (OKS) is a questionnaire used to measure knee pain and knee function, especially in people with:
  Knee arthritis
  Knee injuries
  Before and after knee surgery (like knee replacement)
  It focuses on how knee problems affect daily life.
  What does the test include?
  12 questions
  Each question asks about:
  Knee pain
  Walking
  Standing up
  Climbing stairs
  Night pain
  Daily activities
  The questions usually ask how things have been over the past 4 weeks.
  How is it scored?
  Each question is scored from 0 to 4:
  0 = severe problems
  4 = no problems
  Total score range:
  0 to 48
  How to interpret the score?
  0-19 → Severe knee problems
  20-29 → Moderate knee problems
  30-39 → Mild knee problems
  40-48 → Good knee function
  Higher score = better knee function and less pain
  Why is it used?
  To understand how much knee problems affect daily life
  To measure improvement after treatment or surgery
  To compare patient outcomes in research
SF-12 Physical, and SF-12 Mental scores | From preop to 6 weeks
  What is the SF-12? SF-12 stands for Short Form-12. It has 12 questions about how a person feels and functions in daily life. It's a shorter version of the SF-36 survey and is often used in clinics, research, and public health studies.
  What do P and M mean?
  The SF-12 produces two main scores:
  1. P = Physical Component Summary (PCS)
     This score reflects physical health, including:
     Physical functioning (e.g., ability to do daily activities) Bodily pain General physical health Limitations due to physical problems Higher P (PCS) score → better physical health
  2. M = Mental Component Summary (MCS)
  This score reflects mental and emotional health, including:
  Mood and emotional well-being Stress and anxiety Social functioning Limitations due to emotional problems Higher M (MCS) score → better mental health How are the scores interpreted?
  Scores are usually standardized so that:
  50 = average (based on the general population) Above 50 = better than average Below 50 = worse than average
Timed Up and Go (TUG) test | through study completion, an average of 6 week
  What is the Timed Up and Go (TUG) test?
  The TUG test is a simple physical test used to measure:
  Mobility
  Balance
  Walking ability
  Risk of falling
  It's commonly used in clinics, hospitals, and research, especially for people with muscle, joint, or balance problems.
  How is the test done?
  The person starts sitting in a chair (with armrests).
  On the signal "go," the person:
  Stands up
  Walks 3 meters (about 10 feet)
  Turns around
  Walks back
  Sits down again
  The time is measured in seconds from standing up to sitting back down.
  Assistive devices (like a cane or walker) can be used if normally needed.
  How is it scored?
  The score is the time in seconds.
  Lower time = better mobility
  Common interpretation (may vary slightly):
  < 10 seconds → Normal mobility
  10-19 seconds → Good mobility, mostly independent
  20-29 seconds → Mobility problems, higher fall risk
  ≥ 30 seconds → Severe mobility limitation, very high fall risk
Stair Climb Test (SCT) | through study completion, an average of 6 week
  What is the Stair Climb Test (SCT)?
  The Stair Climb Test is a functional performance test used to assess:
  Lower-limb strength
  Balance and coordination
  Mobility
  Ability to perform daily activities
  It is commonly used in people with knee or hip problems, arthritis, or after lower-limb surgery (such as knee replacement).
  How is the test performed?
  There are a few variations, but the most common method is:
  The person starts standing at the bottom of a staircase.
  On the signal "go," they:
  Climb a set number of stairs (often 9-12 steps)
  Sometimes turn around and come back down (depending on the protocol)
  The time is recorded in seconds.
  * Handrails may be used if needed
  * Assistive devices may be allowed depending on the test rules
  How is it scored?
  The score is the time (in seconds) needed to complete the task.
  Shorter time = better performance
  Some studies also record:
  Time to go up only
  Time to go up and down
  Pain or difficulty during the test
6-minute walk tests | through study completion, an average of 6 week
  The 6MWT is a simple physical fitness test that measures how far a person can walk in 6 minutes.
  It reflects functional exercise capacity-how well someone can perform everyday physical activities.
  It's widely used in people with:
  Heart or lung conditions
  Muscle or joint problems (hip/knee conditions)
  Neurological conditions
  After surgery or rehabilitation
  How is the test performed?
  The person walks back and forth along a flat corridor (usually 20-30 meters long).
  They are instructed to walk as far as possible in 6 minutes at a safe, comfortable pace.
  The person may:
  Slow down
  Stop
  Rest (but the timer keeps running)
  At 6 minutes, the total distance walked is measured (in meters).
  * Normal walking aids may be used
  * Encouragement is usually standardized
  How is it scored?
  The result is the distance walked in 6 minutes (meters).
  Longer distance = better functional capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Functional outcomes and length of stay with early and high-intensity rehabilitation after simultaneous bilateral total knee arthroplasty — https://pubmed.ncbi.nlm.nih.gov/35848009/